CLINICAL TRIAL: NCT02526511
Title: Pilot Study of Renal Neoplasms With Perfusion Magnetic Resonance Imaging
Brief Title: Perfusion Magnetic Resonance Imaging in Diagnosing Patients With Kidney Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, David Foran, PROF-TE-DIR, CINJ-BIOINFORMATICS, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 081407; NCI-2015-00848 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro2013003918 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2015-07-07; First posted 2015-08-18 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Stage I Renal Cell Cancer; Stage II Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnostic (pMRI) (Experimental): Patients undergo DCE, DSC, or ASL pMRI within 30 days of biopsy or surgery. Patients with organ confined tumors selected for active surveillance or surgery and patients with metastatic renal cell carcinoma undergo follow up pMRI at 1-6 months.
  Interventions: Procedure: Arterial Spin Labeling Magnetic Resonance Imaging; Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging; Procedure: Perfusion Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Arterial Spin Labeling Magnetic Resonance Imaging — Undergo arterial spin labeled perfusion magnetic resonance imaging
  Other Names: ARTERIAL SPIN LABELING FUNCTIONAL MRI; Arterial Spin Labeling MRI; ASL; ASL fMRI
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo dynamic contrast-enhanced perfusion magnetic resonance imaging
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Procedure: Dynamic Susceptibility Contrast-Enhanced Magnetic Resonance Imaging — Undergo dynamic susceptibility contrast-enhanced perfusion magnetic resonance imaging
  Other Names: Dynamic Susceptibility Contrast-Enhanced MRI
Procedure: Perfusion Magnetic Resonance Imaging — Undergo perfusion magnetic resonance imaging
  Other Names: magnetic resonance perfusion imaging

SUMMARY:
This pilot clinical trial studies perfusion magnetic resonance imaging in diagnosing patients with kidney tumors. Diagnostic procedures, such as perfusion magnetic resonance imaging, may help find and diagnose kidney tumors and predict and monitor a patient's response to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the utility of perfusion magnetic resonance imaging (pMRI) as a diagnostic biomarker for the prediction of malignant vs. benign organ confined renal masses.

II. To investigate the utility of pMRI as a therapeutic biomarker for monitoring tumor progression in patients undergoing treatment (ablation, surgery, specific systemic treatments such as interleukin 2 (IL-2) or vascular endothelial growth factor [VEGF]/vascular endothelial growth factor receptor [VEGFR]/mechanistic target of rapamycin [mTOR] targeted therapies) or active surveillance for organ confined or metastatic renal tumors.

SECONDARY OBJECTIVES:

I. To investigate the utility of pMRI to predict tumor grade and histologic subtype of organ confined kidney cancers.

OUTLINE:

Patients undergo dynamic contrast enhanced (DCE), dynamic susceptibility contrast (DSC), or arterial spin labeled (ASL) pMRI within 30 days of biopsy or surgery. Patients with organ confined tumors selected for active surveillance or surgery and patients with metastatic renal cell carcinoma undergo follow up pMRI at 1-6 months.

After completion of study, patients are followed up within 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to read, understand, and voluntarily sign an informed consent document
* For patients with organ confined renal tumors to be enrolled, the renal mass must be >= 1 cm in diameter on computed tomography (CT) or magnetic resonance imaging (MRI) and can be any clinical stage T1a-T4 (non-metastatic); a histologic diagnosis is not required for enrollment; the primary imaging site would be kidney
* For patients with metastatic renal tumors to be enrolled, a histologic diagnosis of renal cell carcinoma must exist and any burden of disease >= 1 cm by CT or MRI is acceptable; the metastatic sites may be kidney, intra-abdominal (such as liver), brain, bone, or lymph nodes; lung lesions are NOT eligible because of the motion artifact caused by respiration
* Patients with metastatic disease may have received prior nephrectomy and/or prior systemic therapy (no limit on number); their baseline pMRI would be performed prior to starting a new treatment
* Negative pregnancy test if female of child-bearing age
* Able to undergo contrast enhanced MRI

Exclusion Criteria:

* Severe concurrent disease, infection, or medical co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment
* Severe renal function impairment (estimated glomerular filtration rate [eGFR] < 45 mL/min/1.73 m^2) would make the patient inappropriate for enrollment due to the increased risk of nephrogenic systemic fibrosis (NSF) with higher dose of IV gadolinium-based contrast agents (GBCA) administration
* Women who are pregnant or breastfeeding
* Subjects who are unable to tolerate or are not eligible for MR imaging (claustrophobia, metal implantable devices such as pacemaker, aneurysm clips, etc)
* Subjects with established allergy to IV GBCA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2025-07-28 (Estimated); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
Perfusion MRI outputs | Up to 6 months
  Univariate and multivariate analyses will be performed to look for associations between pMRI outputs and tumor histopathology. The utilization of perfusion MRI as a diagnostic biomarker for tumor grade and histological subtype will be assessed by correlative comparison to histological evaluation by pathology.
Progression free survival | Up to 6 months
  Kaplan-Meier survival curves will be performed to compare groups of patients to assess progression-free survival.
Sensitivity of pMRI | Up to 6 months
  If possible, receiver operating characteristic curves will be created from pMRI data.
Specificity of pMRI | Up to 6 months
  If possible, receiver operating characteristic curves will be created from pMRI data.
Tumor histopathology | Up to 6 months
  Univariate and multivariate analyses will be performed to look for associations between pMRI outputs and tumor histopathology. The utilization of perfusion MRI as a diagnostic biomarker for tumor grade and histological subtype will be assessed by correlative comparison to histological evaluation by pathology.
Progression free survival and/or radiographic tumor evaluation | Up to 6 months
  The utility of pMRI as a therapeutic biomarker for monitoring or predicting treatment response will be assessed by correlative comparison to progression free survival and/or radiographic tumor evaluation by standard of care radiologic imaging modality, such as Response Evaluation Criteria in Solid Tumors.

CONTACTS AND LOCATIONS:
Overall Officials: David Foran, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No